CLINICAL TRIAL: NCT06050317
Title: Sintilimab Plus Chemotherapy and Radiotherapy for Patients With Inoperable Pancreatic Cancer: a Single-arm, Exploratory, Phase II Trial
Brief Title: Sintilimab Combined With Chemotherapy and Radiotherapy in Patients With Inoperable Pancreatic Cancer
Status: Recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Shandong Cancer Hospital and Institute (Other)
Responsible Party: Principal Investigator, Jinbo Yue, Jinbo Yue, Shandong Cancer Hospital and Institute
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: SDZLEC2023-227-02
Record Dates: First submitted 2023-09-17; First posted 2023-09-22 (Actual); Last update posted 2025-07-22 (Actual); Status verified 2025-02

CONDITIONS: Pancreas Cancer
Keywords: Immunothrapy; Chemotherapy; Radiothrapy; Pancreatic cancer
MeSH Terms: conditions — Pancreatic Neoplasms | interventions — sintilimab; Radiation

STUDY DESIGN:
Intervention Model Description: Sintilimab Plus Chemotherapy and Radiotherapy
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (1):
- Sintilimab Plus Chemotherapy and Radiotherapy (Experimental): Sintilimab Plus mFFN or NALIRIFOX and Radiation
  Interventions: Drug: Sintilimab Plus mFFN or NALIRIFOX and Radiation

INTERVENTIONS:
Drug: Sintilimab Plus mFFN or NALIRIFOX and Radiation — Sintilimab Plus mFFN or NALIRIFOX and Radiation
  Other Names: Arm

SUMMARY:
Hypothesis: Survival benefits could be found in Sintilimab plus chemotherapy and radiotherapy in patients with inoperable pancreatic cancer.

DETAILED DESCRIPTION:
Background and aim:

Pancreatic cancer, characterized by its aggressive nature and dismal prognosis, exhibits one of the lowest 5-year survival rates among all solid tumors, standing at a mere 7%. Alarming projections suggest that by the year 2030, it will ascend to become the second leading cause of cancer-related deaths. This dire scenario is further compounded by the stealthy onset of the disease, with an overwhelming 80-85% of patients already presenting with unresectable pancreatic cancer at the time of initial diagnosis.

Clinical trials have endeavored to extend the survival of this challenging patient subset through the administration of chemotherapy or chemoradiotherapy. While these interventions have shown some promise, the overall response rate remains disappointingly low, and patients continue to grapple with a bleak prognosis, often surviving less than a year. This unmet medical need underscores the critical demand for more effective therapeutic modalities in the management of pancreatic cancer, as the lack of viable treatment options remains a primary driver of its high mortality rate.

The traditional therapeutic landscape for unresectable pancreatic cancer primarily relies on single-agent chemotherapy. However, there is a growing realization within the medical community that a paradigm shift toward a multidisciplinary approach is imperative. The crux of achieving long-term survival for pancreatic cancer patients lies in the attainment of a durable anti-tumor response.

Targeted PD-(L)1 immunotherapy, renowned for its ability to induce enduring anti-tumor responses by harnessing the body's own immune system, has yielded remarkable results in various malignancies. Paradoxically, the success of single-agent immunotherapy in pancreatic cancer has been elusive, a phenomenon possibly attributed to the tumor's intrinsic genetic mutations and the hostile, immunosuppressive microenvironment that envelops pancreatic tumors.

Radiation therapy has emerged as a potential ally in this battle against pancreatic cancer. It has been demonstrated to augment the release of tumor-associated antigens, thereby priming the immune system for a more robust response. In response to the resistance encountered with PD-(L)1 monotherapy, researchers have embarked on a journey of preclinical and clinical investigations aimed at validating the combinatorial approach of PD-(L)1 inhibitors alongside chemotherapy and radiation therapy.

The fundamental premise underlying the synergy of radiation and immunotherapy is rooted in the non-invasive initiation of the immune system against tumor cells. Radiation serves as a catalyst, promoting antigen presentation and co-stimulation, culminating in the generation of an immune response targeted at epitopes that had remained concealed within distant metastases. Immune checkpoint inhibitors play a pivotal role in reversing the immunosuppressive effects of the tumor microenvironment, thereby fostering a milieu conducive to anti-tumor immunity.

While the efficacy of this integrative approach remains uncharted territory, current recommendations advocate for a first-line treatment strategy consisting of chemotherapy with optional radiation therapy. Targeted therapy and immunotherapy are not currently included in the initial treatment regimen. Consequently, the primary aim of our study is to explore and elucidate the outcomes of combining Sintilimab with radiation therapy and chemotherapy in the treatment of unresectable pancreatic cancer, offering a glimmer of hope in a landscape fraught with challenges and adversity.

ELIGIBILITY:
Inclusion Criteria:

* ECOG PS 0-1
* Pathological tissue-confirmed unresectable locally advanced pancreatic cancer
* Pancreatic cancer patients who have not received systemic anti-tumor therapy
* Primary pancreatic cancer or at least one measurable lesion specified by RECIST1.1 standards
* A life expectancy of > 3 months
* Blood routine examination: Absolute neutrophil count (ANC) ≥ 1.0 ×109 cells/L, platelets ≥ 75×109 cells/L, hemoglobin ≥ 9.0 g/dl
* AST<2.5 × ULN(Upper Limit of Normal), ALT<2.5 × ULN,creatinine ≤1.5xULN, total bilirubin < ≤1.5 X ULN.

Exclusion Criteria:

* Diagnosed with other malignant diseases other than pancreatic cancer within three years before enrollment
* Patients who are currently participating in interventional clinical research treatment or have received other research drugs or used research devices within four weeks before enrollment
* Patients who have previously received anti-PD-1, anti-PD-L1, or anti-PD-L2 drugs or another drug that stimulates or synergistically inhibits T-cell receptors
* Patients who have received systemic treatment with Chinese patent medicines with anti-tumor indications or drugs with immunomodulatory effects within two weeks before enrollment
* Abnormal results of blood routine examinations and liver and kidney and coagulation tests
* Abnormal function of major organs (14 days before enrollment)
* Women who are pregnant
* Inability of the research subject or authorized legal representative to understand and the willingness to sign a written informed consent document.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 25 (Estimated)
Dates: Start 2023-08-18 (Actual); Primary Completion 2025-08-18 (Estimated); Study Completion 2026-08-18 (Estimated)

PRIMARY OUTCOMES:
PFS | 2 year
  Time from first dose of study drug to first radiographic disease progression or death, whichever occurs first
AE | 2 year
  Advent event rate

SECONDARY OUTCOMES:
Overal response rate | 2 year
  Proportion of subjects with complete response (CR) and partial response (PR) to total subjects; including assessment of irradiated lesions and non-irradiated lesions
Overall survival | 2 year
  The time from the start of treatment to death
Disease control rate | 2 year
  Proportion of total subjects defined as complete response (CR), partial response (PR), and stable disease (SD)
Duration of response | 2 year
  The time from when the tumor is first evaluated as CR or PR to when the tumor is first evaluated as PD (Progressive Disease) or death from any cause

CONTACTS AND LOCATIONS:
Overall Officials: Jinbo Yue, dorctor, Principal Investigator — Shandong Cancer Hospital and Institute
Locations (1):
- Department of Radiation Oncology, Shandong Cancer Hospital and Institute, Jinan, Shandong, China

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Ilic M, Ilic I. Epidemiology of pancreatic cancer. World J Gastroenterol. 2016 Nov 28;22(44):9694-9705. doi: 10.3748/wjg.v22.i44.9694. PMID 27956793
- [Background] Rahib L, Smith BD, Aizenberg R, Rosenzweig AB, Fleshman JM, Matrisian LM. Projecting cancer incidence and deaths to 2030: the unexpected burden of thyroid, liver, and pancreas cancers in the United States. Cancer Res. 2014 Jun 1;74(11):2913-21. doi: 10.1158/0008-5472.CAN-14-0155. PMID 24840647
- [Background] Strohl MP, Raigani S, Ammori JB, Hardacre JM, Kim JA. Surgery for Localized Pancreatic Cancer: The Trend Is Not Improving. Pancreas. 2016 May-Jun;45(5):687-93. doi: 10.1097/MPA.0000000000000511. PMID 26491905
- [Background] Conroy T, Desseigne F, Ychou M, Bouche O, Guimbaud R, Becouarn Y, Adenis A, Raoul JL, Gourgou-Bourgade S, de la Fouchardiere C, Bennouna J, Bachet JB, Khemissa-Akouz F, Pere-Verge D, Delbaldo C, Assenat E, Chauffert B, Michel P, Montoto-Grillot C, Ducreux M; Groupe Tumeurs Digestives of Unicancer; PRODIGE Intergroup. FOLFIRINOX versus gemcitabine for metastatic pancreatic cancer. N Engl J Med. 2011 May 12;364(19):1817-25. doi: 10.1056/NEJMoa1011923. PMID 21561347
- [Background] Burris HA 3rd, Moore MJ, Andersen J, Green MR, Rothenberg ML, Modiano MR, Cripps MC, Portenoy RK, Storniolo AM, Tarassoff P, Nelson R, Dorr FA, Stephens CD, Von Hoff DD. Improvements in survival and clinical benefit with gemcitabine as first-line therapy for patients with advanced pancreas cancer: a randomized trial. J Clin Oncol. 1997 Jun;15(6):2403-13. doi: 10.1200/JCO.1997.15.6.2403. PMID 9196156
- [Background] Von Hoff DD, Ervin T, Arena FP, Chiorean EG, Infante J, Moore M, Seay T, Tjulandin SA, Ma WW, Saleh MN, Harris M, Reni M, Dowden S, Laheru D, Bahary N, Ramanathan RK, Tabernero J, Hidalgo M, Goldstein D, Van Cutsem E, Wei X, Iglesias J, Renschler MF. Increased survival in pancreatic cancer with nab-paclitaxel plus gemcitabine. N Engl J Med. 2013 Oct 31;369(18):1691-703. doi: 10.1056/NEJMoa1304369. Epub 2013 Oct 16. PMID 24131140
- [Background] Fukumura D, Jain RK. Tumor microvasculature and microenvironment: targets for anti-angiogenesis and normalization. Microvasc Res. 2007 Sep-Nov;74(2-3):72-84. doi: 10.1016/j.mvr.2007.05.003. Epub 2007 May 18. PMID 17560615
- [Background] Badiyan SN, Molitoris JK, Chuong MD, Regine WF, Kaiser A. The Role of Radiation Therapy for Pancreatic Cancer in the Adjuvant and Neoadjuvant Settings. Surg Oncol Clin N Am. 2017 Jul;26(3):431-453. doi: 10.1016/j.soc.2017.01.012. Epub 2017 May 11. PMID 28576181
- [Background] Auclin E, Marthey L, Abdallah R, Mas L, Francois E, Saint A, Cunha AS, Vienot A, Lecomte T, Hautefeuille V, de La Fouchardiere C, Sarabi M, Ksontini F, Forestier J, Coriat R, Fabiano E, Leroy F, Williet N, Bachet JB, Tougeron D, Taieb J. Role of FOLFIRINOX and chemoradiotherapy in locally advanced and borderline resectable pancreatic adenocarcinoma: update of the AGEO cohort. Br J Cancer. 2021 Jun;124(12):1941-1948. doi: 10.1038/s41416-021-01341-w. Epub 2021 Mar 26. PMID 33772154
- [Background] Loehrer PJ Sr, Feng Y, Cardenes H, Wagner L, Brell JM, Cella D, Flynn P, Ramanathan RK, Crane CH, Alberts SR, Benson AB 3rd. Gemcitabine alone versus gemcitabine plus radiotherapy in patients with locally advanced pancreatic cancer: an Eastern Cooperative Oncology Group trial. J Clin Oncol. 2011 Nov 1;29(31):4105-12. doi: 10.1200/JCO.2011.34.8904. Epub 2011 Oct 3. PMID 21969502
- [Background] Chauffert B, Mornex F, Bonnetain F, Rougier P, Mariette C, Bouche O, Bosset JF, Aparicio T, Mineur L, Azzedine A, Hammel P, Butel J, Stremsdoerfer N, Maingon P, Bedenne L. Phase III trial comparing intensive induction chemoradiotherapy (60 Gy, infusional 5-FU and intermittent cisplatin) followed by maintenance gemcitabine with gemcitabine alone for locally advanced unresectable pancreatic cancer. Definitive results of the 2000-01 FFCD/SFRO study. Ann Oncol. 2008 Sep;19(9):1592-9. doi: 10.1093/annonc/mdn281. Epub 2008 May 7. PMID 18467316
- [Background] Hammel P, Huguet F, van Laethem JL, Goldstein D, Glimelius B, Artru P, Borbath I, Bouche O, Shannon J, Andre T, Mineur L, Chibaudel B, Bonnetain F, Louvet C; LAP07 Trial Group. Effect of Chemoradiotherapy vs Chemotherapy on Survival in Patients With Locally Advanced Pancreatic Cancer Controlled After 4 Months of Gemcitabine With or Without Erlotinib: The LAP07 Randomized Clinical Trial. JAMA. 2016 May 3;315(17):1844-53. doi: 10.1001/jama.2016.4324. PMID 27139057
- [Background] Radiation therapy combined with Adriamycin or 5-fluorouracil for the treatment of locally unresectable pancreatic carcinoma. Gastrointestinal Tumor Study Group. Cancer. 1985 Dec 1;56(11):2563-8. doi: 10.1002/1097-0142(19851201)56:113.0.co;2-0. PMID 2864997
- [Background] de Geus SWL, Eskander MF, Kasumova GG, Ng SC, Kent TS, Mancias JD, Callery MP, Mahadevan A, Tseng JF. Stereotactic body radiotherapy for unresected pancreatic cancer: A nationwide review. Cancer. 2017 Nov 1;123(21):4158-4167. doi: 10.1002/cncr.30856. Epub 2017 Jul 14. PMID 28708929
- [Background] Tchelebi LT, Lehrer EJ, Trifiletti DM, Sharma NK, Gusani NJ, Crane CH, Zaorsky NG. Conventionally fractionated radiation therapy versus stereotactic body radiation therapy for locally advanced pancreatic cancer (CRiSP): An international systematic review and meta-analysis. Cancer. 2020 May 15;126(10):2120-2131. doi: 10.1002/cncr.32756. Epub 2020 Mar 3. PMID 32125712
- [Background] Zhong J, Patel K, Switchenko J, Cassidy RJ, Hall WA, Gillespie T, Patel PR, Kooby D, Landry J. Outcomes for patients with locally advanced pancreatic adenocarcinoma treated with stereotactic body radiation therapy versus conventionally fractionated radiation. Cancer. 2017 Sep 15;123(18):3486-3493. doi: 10.1002/cncr.30706. Epub 2017 May 10. PMID 28493288
- [Background] Hewitt DB, Nissen N, Hatoum H, Musher B, Seng J, Coveler AL, Al-Rajabi R, Yeo CJ, Leiby B, Banks J, Balducci L, Vaccaro G, LoConte N, George TJ, Brenner W, Elquza E, Vahanian N, Rossi G, Kennedy E, Link C, Lavu H. A Phase 3 Randomized Clinical Trial of Chemotherapy With or Without Algenpantucel-L (HyperAcute-Pancreas) Immunotherapy in Subjects With Borderline Resectable or Locally Advanced Unresectable Pancreatic Cancer. Ann Surg. 2022 Jan 1;275(1):45-53. doi: 10.1097/SLA.0000000000004669. PMID 33630475
- [Background] Chen IM, Donia M, Chamberlain CA, Jensen AWP, Draghi A, Theile S, Madsen K, Hasselby JP, Toxvaerd A, Hogdall E, Lorentzen T, Wilken EE, Geertsen P, Svane IM, Johansen JS, Nielsen D. Phase 2 study of ipilimumab, nivolumab, and tocilizumab combined with stereotactic body radiotherapy in patients with refractory pancreatic cancer (TRIPLE-R). Eur J Cancer. 2023 Feb;180:125-133. doi: 10.1016/j.ejca.2022.11.035. Epub 2022 Dec 10. PMID 36592507
- [Background] Ahmad G, Mackenzie GG, Egan J, Amiji MM. DHA-SBT-1214 Taxoid Nanoemulsion and Anti-PD-L1 Antibody Combination Therapy Enhances Antitumor Efficacy in a Syngeneic Pancreatic Adenocarcinoma Model. Mol Cancer Ther. 2019 Nov;18(11):1961-1972. doi: 10.1158/1535-7163.MCT-18-1046. Epub 2019 Aug 22. PMID 31439714
- [Background] Weiss GJ, Blaydorn L, Beck J, Bornemann-Kolatzki K, Urnovitz H, Schutz E, Khemka V. Phase Ib/II study of gemcitabine, nab-paclitaxel, and pembrolizumab in metastatic pancreatic adenocarcinoma. Invest New Drugs. 2018 Feb;36(1):96-102. doi: 10.1007/s10637-017-0525-1. Epub 2017 Nov 8. PMID 29119276
- [Background] Padron LJ, Maurer DM, O'Hara MH, O'Reilly EM, Wolff RA, Wainberg ZA, Ko AH, Fisher G, Rahma O, Lyman JP, Cabanski CR, Yu JX, Pfeiffer SM, Spasic M, Xu J, Gherardini PF, Karakunnel J, Mick R, Alanio C, Byrne KT, Hollmann TJ, Moore JS, Jones DD, Tognetti M, Chen RO, Yang X, Salvador L, Wherry EJ, Dugan U, O'Donnell-Tormey J, Butterfield LH, Hubbard-Lucey VM, Ibrahim R, Fairchild J, Bucktrout S, LaVallee TM, Vonderheide RH. Sotigalimab and/or nivolumab with chemotherapy in first-line metastatic pancreatic cancer: clinical and immunologic analyses from the randomized phase 2 PRINCE trial. Nat Med. 2022 Jun;28(6):1167-1177. doi: 10.1038/s41591-022-01829-9. Epub 2022 Jun 3. PMID 35662283
- [Background] Zhu X, Cao Y, Liu W, Ju X, Zhao X, Jiang L, Ye Y, Jin G, Zhang H. Stereotactic body radiotherapy plus pembrolizumab and trametinib versus stereotactic body radiotherapy plus gemcitabine for locally recurrent pancreatic cancer after surgical resection: an open-label, randomised, controlled, phase 2 trial. Lancet Oncol. 2021 Aug;22(8):1093-1102. doi: 10.1016/S1470-2045(21)00286-2. Epub 2021 Jul 5. PMID 34237249
- [Background] Chen IM, Johansen JS, Theile S, Hjaltelin JX, Novitski SI, Brunak S, Hasselby JP, Willemoe GL, Lorentzen T, Madsen K, Jensen BV, Wilken EE, Geertsen P, Behrens C, Nolsoe C, Hermann KL, Svane IM, Nielsen D. Randomized Phase II Study of Nivolumab With or Without Ipilimumab Combined With Stereotactic Body Radiotherapy for Refractory Metastatic Pancreatic Cancer (CheckPAC). J Clin Oncol. 2022 Sep 20;40(27):3180-3189. doi: 10.1200/JCO.21.02511. Epub 2022 Apr 27. PMID 35476508